CLINICAL TRIAL: NCT03748030
Title: Assessing Acute Cardiac Inflammation After Left-Sided Breast Cancer Radiotherapy With Hybrid PET/MRI
Brief Title: Hybrid PET/MR Imaging of Acute Cardiac Inflammation After Left-Sided Breast Cancer Radiotherapy
Acronym: RICT-BREAST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 112991
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Left-Sided Breast Cancer; Radiation Toxicity
MeSH Terms: conditions — Unilateral Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Confirmed Left-Sided Breast Cancer: T1/T2 N0, T1/T2 N1, T3/T4 and/or N2/N3 Left-Sided Breast Cancer Patients receiving standard radiation therapy will receive PET/MRI, ECG/EKG, and bloodwork before, within a month, and within a year post treatment.
  Interventions: Radiation: Confirmed Left-Sided Breast Cancer

INTERVENTIONS:
Radiation: Confirmed Left-Sided Breast Cancer — Left-Sided Patients will receive standard radiation therapy, including 42.5 Gy in 16 fractions or 50 Gy in 25 fractions.

SUMMARY:
Radiation therapy (RT) of the breast is a critical component of modern breast cancer treatment. RT treatments have led to improved local control and overall survival of breast cancer patients. However, the incidence of radiation induced harmful effects is increasing in these patients. This is because in delivering RT, it is difficult to completely avoid surrounding non-cancerous normal tissue, including the heart. The main concern here is that radiation induced effects on the heart may lead to an increased risk of cardiovascular disease later in a patient's life, potentially many years after radiation. Despite methods that can detect alterations in blood flow one to two years following radiotherapy, knowledge of early radiation effects to the heart is still limited. A previous animal experiment performed by our group involved delivering a radiation dose to the heart in a manner similar to the way a heart would be exposed, during radiotherapy for a cancer involving the left breast. Taking several images over the months following radiation with a new imaging technique, hybrid PET/MRI, has suggested an increase in inflammation can be detected as early as one-week following irradiation and may be the triggering event for cardiac disease seen in women 10-15 years after radiotherapy. The investigators propose a pilot study where 15 left-sided breast cancer patients undergoing radiotherapy will be imaged before, as well as one week and one-year post radiotherapy with our hybrid PET/MRI scanner. Areas of inflammation, changes in blood flow, and scar formation within the heart, will be measured by looking at the difference between images that are taken after radiation treatment to the images taken before treatment. The expectation is that any areas of the heart that show detectable differences in the images will be directly related to how much radiation was deposited in those areas. The information gained from this pilot study which will correlate the amount of radiation administered to the degree and extent of injury will help aid in the design of new treatment strategies, that can hopefully decrease or eliminate inadvertent heart damage, thereby, improving the quality of life for breast cancer patients.

DETAILED DESCRIPTION:
Goals: The overall goal of this study is to identify the presence of acute low-dose radiation induced cardiac toxicity, including inflammation, in left-sided breast cancer patients undergoing radiotherapy using hybrid positron emission tomography (PET) and magnetic resonance imaging (MRI).

Methodology: A imaging pilot study composed of 15 left-sided breast cancer patients receiving standard radiotherapy is proposed. Patients will be imaged at baseline, within the first month post radiotherapy, and within the first-year post radiotherapy using a hybrid 3T-PET/MRI system (Biograph mMR, Siemens Healthcare). The PET imaging protocol is designed to assess changes in both myocardial perfusion and inflammation. The MR imaging protocol, acquired simultaneously, will be used to identify heart volume, wall motion, mature fibrosis or scar.

Outcome: The findings of this studies will validate the utility of hybrid PET/MRI to detect early inflammatory response, changes in myocardial perfusion, and heart function as a function of radiation dose in a human breast cancer population. This will allow consideration of new techniques to minimize or eliminate heart complications to future cancer patients and provide a non-invasive technique to serially image patients post radiotherapy and to investigate the effect of new interventions. Success of this study will stem from a unique collaboration of Radiation Oncologists, Medical Physicists, Imaging Scientists, and Cardiologists.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Ability to provide informed consent
* Histologically evidence of left-sided breast cancer where potentially curative treatment is planned
* T1/T2 N0, T1/T2 N1, T3/T4 and/or N2/N3 according to Tumor-Node-Metastases (TNM) staging criteria
* All patients to receive prescription dose according to current London Regional Cance Program (LRCP) standards
* No prior RT to the thorax
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 within one month of accrual
* Satisfactory pulmonary function as determined by the treating radiation oncologist
* Expected lifespan at least 1 year
* Negative pregnancy test within one month of accrual if woman is premenopausal

Exclusion Criteria:

* No current or recurring atrial fibrillation
* Previous coronary bypass surgery
* Patients with severe reversible airways obstruction
* Patients with acute coronary syndrome (STEMI/non-STEMI and unstable angina)
* Atrioventricular block without pacemaker
* Patients who are renal insufficient (eGFR <40)
* Patients with asthma
* Allergy to gadolinium for scans using contrast; will be eligible for non-contrast scans.
* Other contraindications to gadolinium contrast media as determined by the research team.
* Relative contraindications to PET (e.g. uncontrolled diabetes, claustrophobia, inability to be still for 60 minutes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ultimately, the sample size was based upon practical considerations and that 15 breast cancer patients could be accrued relatively easily from new patient clinics, while sufficiently providing enough evidence to validate the imaging techniques to be used as a non-invasive measure for future clinical trials aimed at reducing or mitigating radiation-induced cardiac toxicity.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Imaging Biomarkers of acute cardiac inflammation | one month
  18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG)-PET imaging to detect increase in cardiac inflammation compared to baseline with corresponding blood markers (Erythrocyte Sedimentation Rate (ESR), high sensitivity C-reactive protein, and troponin levels in blood (inflammation)).
Detection of Imaging Biomarkers of late cardiac inflammation | one year
  FDG-PET imaging to detect increase in cardiac inflammation compared to baseline with corresponding blood markers (Erythrocyte Sedimentation Rate (ESR), high sensitivity C-reactive protein, and troponin levels in blood (inflammation)).
Detection of Imaging Biomarkers of acute cardiac perfusion changes | one month
  N-13 Ammonia PET imaging to detect changes in acute cardiac perfusion changes compared to baseline.
Detection of Imaging Biomarkers of late cardiac perfusion changes | one year
  N-13 Ammonia PET imaging to detect changes in late cardiac perfusion changes
Detection of cardiac fibrosis | one year
  Gadolinium Enhanced MR imaging to detect cardiac fibrosis compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Gaede, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No